CLINICAL TRIAL: NCT06992622
Title: Zhejiang Adolescent Spine and Vision Health Cohort: A Longitudinal Database Analysis
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Xiangyang Wang, M.D., Chief physician, Doctorial supervisor, Second Affiliated Hospital of Wenzhou Medical University
Other Study IDs: SAHoWMU-CR2025-08-220
Record Dates: First submitted 2025-05-08; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Scoliosis Idiopathic; Myopia; Vision Disorders
Keywords: Adolescent idiopathic scoliosis; Longitudinal progression; Spine-vision comorbidity
MeSH Terms: conditions — Myopia; Vision Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IS with Myopia: diopathic scoliosis with untreated myopia
- IS without Myopia: diopathic scoliosis without myopia

SUMMARY:
The aim of study: 1. To investigate the prevalence of scoliosis, other spinal deformities, myopia, and visual impairments in adolescents (aged 6-18) in Zhejiang Province.

2.To track 8-year dynamic changes in spinal curvature and analyze associations between scoliosis, vision disorders, and potential risk factors.

3.To deliver scoliosis health education during screenings.

4.To mitigate scoliosis progression through early detection and intervention.

DETAILED DESCRIPTION:
Scoliosis is the most common pediatric musculoskeletal disorder, affecting up to 4% of otherwise healthy children worldwide. Approximately 80-90% of cases are idiopathic scoliosis (IS), predominantly emerging during adolescence. While mild IS often causes no symptoms, moderate cases may lead to spinal deformity and mild respiratory dysfunction, with severe cases potentially resulting in cardiopulmonary compromise or even paralysis.

Despite extensive research exploring potential causes - including genetic, neuroendocrine, skeletal, muscular, postural, biomechanical and lifestyle factors - the underlying mechanisms of IS remain unclear. Bracing currently stands as the only proven conservative treatment to slow progression, yet 20-30% of braced patients still require eventual surgical correction. Adolescence represents both a critical window for rapid curve progression and the optimal period for effective intervention. Early screening has been demonstrated to significantly improve outcomes, highlighting the importance of preventive strategies during this developmental stage.

Recent studies across various populations have reported scoliosis prevalence rates ranging from 0.27% to 3.5%, with notable regional variations:

Singaporean studies found rates between 0.27%-2.49%

Greek research reported 1.7% prevalence

Large-scale US screening showed 0.9% prevalence

Chinese studies documented rates from 1.07% (Guangzhou) to 3.5% (Hong Kong)

Most existing research has been cross-sectional in design, lacking prospective data on curve progression patterns and associated risk factors.

This prospective cohort study aims to:1. To investigate the prevalence of scoliosis, other spinal deformities, myopia, and visual impairments in adolescents (aged 6-18) in Zhejiang Province.

2.To track 8-year dynamic changes in spinal curvature and analyze associations between scoliosis, vision disorders, and potential risk factors.

3.To deliver scoliosis health education during screenings.

4.To mitigate scoliosis progression through early detection and intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic scoliosis at their first clinic visit
* Skeletally immature (Risser Sign 0-3)
* Cobb angle between 11-40 degrees
* Age between 6 and 17

Exclusion Criteria:

* • Patients with scoliosis other than idiopathic, or with other musculoskeletal or neurodevelopmental conditions that might be responsible for the scoliosis

  * History of previous spine surgery or spinal injury
  * Tumor or malignant tumor in the spine
  * Leg length discrepancy more than 20 mm
  * Previous diagnosis or treatment of SDB more than 6 months ago
  * Plans to relocate within the next 24 months

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Adolescents participating in the Zhejiang Adolescent Spine and Vision Health Screening Program, China
Sampling Method: Non-Probability Sample
Enrollment: 73000 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2032-09-30 (Estimated); Study Completion 2032-12-30 (Estimated)

PRIMARY OUTCOMES:
Scoliosis Curve Angle | Baseline, 24 months (±1 month), and 48 months (±1 month) after enrollment; data will be analyzed through study completion, up to 96 months.]
  A long standard standing whole spine radiograph will be used for measuring curve size in terms of Cobb angle according to the standard Cobb method
Angle of Trunk Rotation | Baseline, 24 months (±1 month), and 48 months (±1 month) after enrollment; data will be analyzed through study completion, up to 96 months.]
  In addition to spinal x-rays, a Scoliometer can also help monitor curve progression. The Scoliometer is an inclinometer that measures the asymmetries between the sides of the trunk by measuring axial rotation in degrees. Numerous studies have found a high correlation between trunk axial rotation (ATR) values and the Cobb angles.

SECONDARY OUTCOMES:
Cycloplegic Mean Spherical Equivalent (MSE) for Myopia Diagnosis | Baseline and every 24 months (±1 month) until study completion, up to 96 months.
  MSE (diopters) will be calculated as [sphere + ½ cylinder] using autorefraction (Topcon KR-800) under cycloplegia (1% cyclopentolate). Myopia is defined as MSE ≤-0.50D. Triplicate measurements will be averaged per eye.
Daily Near-Work Duration (UVD) Assessed by 30-Minute Block Questionnaire | Baseline, 24 months (±1 month), and 48 months (±1 month) after enrollment; data will be analyzed through study completion, up to 96 months.
  Daily near-work activities (reading/digital screen use) will be recorded through the validated 20-item Near-Vision Activity Questionnaire (NVAQ). Total daily UVD will be calculated by summing 30-minute activity blocks (maximum 16 blocks/day).
Axial Length (AL) Growth Rate Measured by Swept-Source OCT | Baseline, 24 months (±1 month), and 48 months (±1 month) after enrollment; data will be analyzed through study completion, up to 96 months.
  AL (mm) will be measured using swept-source optical coherence tomography (Topcon Triton Plus). Annualized growth rates (mm/year) will be calculated by linear regression of AL against time between baseline and each follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangyang Wang, Study Chair — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang 325000, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided